CLINICAL TRIAL: NCT00065234
Title: Acupuncture to Prevent Postoperative Paralytic Ileus
Brief Title: Acupuncture to Prevent Postoperative Bowel Paralysis (Paralytic Ileus)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21AT001065-01A1 (NIH); ChiangJ
Record Dates: First submitted 2003-07-18; First posted 2003-07-22 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Ileus; Neoplasms
Keywords: Colostomy; Ileostomy
MeSH Terms: conditions — Ileus; Neoplasms | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this study is to determine if acupuncture is effective in preventing prolonged postoperative paralysis of the gastrointestinal tract among patients undergoing colostomy/ileostomy closure.

ELIGIBILITY:
Inclusion Criteria:

* Previous surgical cancer treatment with ileostomy/colostomy, now scheduled for closure
* Hospital admission must be same day as surgery

Exclusion Criteria:

* Incapacitating disease
* Concurrent herbal or laxative use
* Use of Heparin or Coumadin
* Upper or lower extremity deformities
* Chronic constipation prior to cancer diagnosis
* History of cerebrovascular accident or spinal cord injury
* Chronic pain that has been treated with any form of major opioid or weak opioids (=/> 30mg/24 hours)
* Pacemaker or metal implants
* Concurrent alternative medicine/herbal use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-09; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S Chiang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States